CLINICAL TRIAL: NCT04334902
Title: An Open Label, Multicenter, Retrospective, Pivotal Trial to Evaluate the Efficacy of Clinical Decision Support System-mPDia for Neurodegenerative Parkinsonism Using MRI Images
Brief Title: Evaluation of Clinical Decision Support System-mPDia for Neurodegenerative Parkinsonism Using MRI Images
Status: Completed | Type: Observational
Sponsor: Heuron Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HR-MPD-01
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Diagnoses Disease
Keywords: Neurodegenerative Parkinsonism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abnormal: The person who visits parkinsonism symptoms and has been diagnosed with neurodegenerative parkinsonism
  Interventions: Device: mPDia
- Normal: The person who visits parkinsonism symptoms but is not or is normal for neurodegenerative parkinsonism
  Interventions: Device: mPDia

INTERVENTIONS:
Device: mPDia — Clinical decision support system for diagnosing neurodegenerative parkinsonism

SUMMARY:
mPDia is a software that has been pre-learned based on a neurodegenerative parkinsonism diagnosis model using Nigrosome 1 MRI images, and clinical decision support system for diagnosing neurodegenerative parkinsonism by automatically analyzing Nigrosome 1 MRI images by assisting the medical team.

The specific aims of this study are to evaluate efficacy of mPDia for neurodegenerative Parkinsonism compared to the sensitivity and specificity levels of 18F FP-CIT PET/CT which is currently used to diagnose neurodegenerative parkinsonism.

ELIGIBILITY:
Inclusion Criteria(Normal cohort):

* Adults over 19 years old
* 3T nigrosome 1 MRI acquired
* 18F FP-CIT PET/CT are confirmed to be normal
* The person who visits parkinsonism symptoms but is not or is normal for neurodegenerative parkinsonism

Inclusion Criteria(Abnormal cohort):

* Adults over 19 years old
* 3T nigrosome 1 MRI acquired
* 18F FP-CIT PET/CT are confirmed to be abnormal
* The person who visits parkinsonism symptoms and has been diagnosed with neurodegenerative parkinsonism

Exclusion Criteria:

* Patients with other brain diseases except parkinsonism
* Who have anatomical abnormality in MRIs etc.
* Who have other causes of tremor(e.g., thyroid disease)
* Patients with lesion in basal ganglia(e.g., vascular parkinsonism, hydrocephalus and Wilson's disease)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (1) Adults over 19 years old (2) 3T nigrosome 1 MRI acquired (3) 18F FP-CIT PET/CT are confirmed to be normal(normal cohort) or abnormal(abnormal cohort)
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: YoungHee Sung, M.D, Ph.D, Principal Investigator — Gachon University Gil Medical Center
Locations (10):
- South Korea (10):
  - Cha Medical Center, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - KyungHee University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The data will be collected retrospectively from person whose past 3T nigrosome 1 MRI image, 18F FP-CIT PET/CT image, image interpretation, and neurologic exam results are confirmed by medical records, and those whose diagnosis as neurodegenerative Parkinsonism is confirmed. Data collecting must be executed following therandom collection. Only the verified researcher who is registered in this study will have access to medical records.
Pre-assignment Details: At each Institution, participants who met all inclusion and exclusion criteria for this study were randomly selected up to the target number of participants. Based on the medical record diagnosis of neurodegenerative parkinsonism, participants were classified into the normal group or the patient group. The data from the randomly selected participants were used for diagnostic evaluation.
Groups:
- Normal: The person who presented with parkinsonism symptoms but were determined not to have neurodegenerative parkinsonism.
Period: Overall Study
Arm/Group | Abnormal | Normal
Started | 159 | 62
Completed | 158 | 60
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Of the 221 cases(patient group 159 cases, normal group 62 cases) enrolled in this clinical trial, 218 cases(patient group 158 cases-5056 images, normal group 60 cases-1920 images) who completed the trial according to the clinical trial protocol were used as data for efficacy assessment, excluding 3 people (1.36%) dropped out. In the case of demographic information and basic data, the analysis was conducted with the corresponding data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abnormal | Normal | Total
Number analyzed (Participants) | 158 | 60 | 218
Sex: Female, Male [Count of Participants; unit: Participants] — For the demographic information checked at visit 1, in the case of age, descriptive statistics (number, mean, standard deviation, median, minimum, maximum) were presented as continuous variables, and in the case of sex, frequency and percentage (%) were presented as categorical variables Population: Since this clinical trial is not a parallel design comparing two groups, comparative analysis of basic data and test results between the normal group and the patient group was not conducted.
  Participants
    Female | 83 | 36 | 119
    Male | 75 | 24 | 99
Age, Continuous [Mean (Standard Deviation); unit: year] — The mean age of the enrolled cases was 66.54±9.93 years, and subjects from 37 to 90 years old participated, and the mean age of the patient group was 65.85±10.50 years, and the mean age of the normal group was 68.35±8.04 years.
  year | 65.85 (10.50) | 68.35 (8.04) | 66.54 (9.93)
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of mPDia for the Diagnosis of Neurodegenerative Parkinsonism
Description: Sensitivity of mPDia in diagnosing neurodegenerative parkinsonism, based on comparison with the golden standard (final clinical diagnosis determined by specialist groups).
  Sensitivity was calculated as TP/(TP+FN) Sensitivity: 100 x True positive(TP)/ [True positive(TP) + False negative(FN)] (%)
Time Frame: At Visit 2 (within 4 weeks after Visit 1)
Population: Sensitivity is calculated only in the Abnormal group (patients diagnosed with neurodegenerative parkinsonism).
  The Normal group is not applicable for this analysis, therefore the number of participants analyzed is recorded as 0.
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Abnormal | Normal
Number analyzed (Participants) | 158 | 0
percentage | 94.30 [90.69 to 97.92] |

2. Primary Outcome: Specificity of mPDia for the Diagnosis of Neurodegenerative Parkinsonism
Description: Specificity of mPDia in diagnosing neurodegenerative parkinsonism, based on comparison with the golden standard (final clinical diagnosis determined by specialist groups).
  Specificity was calculated as True Negative / (True Negative + False Positive) Specificity: 100 x True negative(TN)/[False positive(FP) + True negative(TN)] (%)
Time Frame: At Visit 2 (within 4 weeks after Visit 1)
Population: Specificity is calculated only in the Normal group (participants without neurodegenerative parkinsonism).
  The Abnormal group is not applicable for this analysis, therefore the number of participants analyzed is recorded as 0.
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Abnormal | Normal
Number analyzed (Participants) | 0 | 60
percentage |  | 91.67 [84.67 to 98.66]

ADVERSE EVENTS:
Time Frame: Not Applilcable(Retrospective Study)
Description: All-Cause Mortality, Serious Adverse Events, and Other (Non-Serious) Adverse Events were not monitored or assessed in this study.
Arm/Group | Abnormal | Normal
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT04334902/Prot_SAP_000.pdf